CLINICAL TRIAL: NCT00948181
Title: Evaluation of Stress Hormone Concentration During the Resection of Pheochromocytoma. Comparison of Surgeon - Anesthesiologist - Patient
Brief Title: Evaluation of Plasma Catecholamine Concentration During Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kliniken Essen-Mitte (Other)
Collaborators: Universität Duisburg-Essen (Other)
Responsible Party: Prof. Dr. Harald Groeben, Kliniken Essen-Mitte
Other Study IDs: 2009061
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2009-07

CONDITIONS: Stress
Keywords: Epinephrine, Norepinephrine, normetanephrine; Catecholamine concentrations during surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood will be drawn from the surgeon, anesthesiologist and from 8 patients to determine plasma catecholamine concentrations. Only plasma will be used for measurements.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Surgeon: To detect the degree of intraoperative stress, venous blod will be drawn from one surgeon during 8 pheochromocytoma resections.
- Anesthesiologist: To detect the degree of intraoperative stress, venous blood will be drawn from one anesthesiologist during 8 pheochromocytoma resections.
- Patients with pheochromocytoma: Venous blood will be drawn from 8 patients with pheochromocytoma during tumor resection.

SUMMARY:
Stress during surgery leads to significant increase in plasma catecholamine concentrations in surgeons, anesthesiologists, and patients.

DETAILED DESCRIPTION:
Hypothesis: Resection of pheochromocytomas can lead to more than normal stress in surgeons and because of abrupt hemodynamic changes in patients as well in anesthesiologists. Measurements of catecholamine concentrations at baseline, prior to surgery during and after surgery, are to be performed to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria: Patients with pheochromocytoma (Older than 18 years) -

Exclusion Criteria: Patients younger than 18 years. Conservative treatment.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of 8 patients with pheochromocytoma scheduled for tumor resection, one surgeon (with the experience of more than 50 pheochromocytoma resections) and one anesthesiologist (with the experience of more than 50 pheochromocytoma resections).
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-07 (Estimated); Study Completion 2010-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Harald Groeben, M.D., Principal Investigator — Kliniken Essen-Mitte
Locations (1):
- Prof. Dr. Harald Groeben, Essen, Germany

REFERENCES:
- [Background] Unger N, Pitt C, Schmidt IL, Walz MK, Schmid KW, Philipp T, Mann K, Petersenn S. Diagnostic value of various biochemical parameters for the diagnosis of pheochromocytoma in patients with adrenal mass. Eur J Endocrinol. 2006 Mar;154(3):409-17. doi: 10.1530/eje.1.02097. PMID 16498054
- [Background] Schuttler J, Westhofen P, Kania U, Ihmsen H, Kammerecker S, Hirner A. [Quantitative assessment of catecholamine secretion as a rational principle of anesthesia management in pheochromocytoma surgery]. Anasthesiol Intensivmed Notfallmed Schmerzther. 1995 Oct;30(6):341-9. doi: 10.1055/s-2007-996507. German. PMID 8541435